CLINICAL TRIAL: NCT01759368
Title: Heart at Home- Remote Patient Monitoring in the Care of Heart Failure Patients
Brief Title: Heart at Home- a Self-care Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VTT Technical Research Centre of Finland (Other)
Collaborators: Helsinki University Central Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HUSHAH
Record Dates: First submitted 2012-12-20; First posted 2013-01-03 (Estimated); Results first posted 2014-09-17 (Estimated); Last update posted 2014-09-17 (Estimated); Status verified 2014-09

CONDITIONS: Heart Failure
Keywords: self-care, heart failure, telemonitoring, health care utilization
MeSH Terms: conditions — Heart Failure; Patient Acceptance of Health Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Telemonitoring assisted self-care (Active Comparator): Telemonitoring group was given a home-care package including a weight scale, a blood pressure meter, a mobile phone and self-care instructions. The measurements taken at home to be uploaded were: diastolic and systolic blood pressure, pulse, body weight and an assessment of symptoms. The symptom assessment concerned the patient's feelings of dizziness, dyspnea, palpitation, weakness and, oedema. Patients were also asked to evaluate their overall condition- whether their condition had deteriorated, improved or remained unchanged. The patients were advised to carry out and report the measurements together with the self-assessment once a week. The responsible nurse followed patients' status and the data once a week or more frequently if needed. Based on the reported measurements, the nurse could invite the patient for a control visit. In case a patient did not make self-measurements as planned , the nurse contacted the patient and reminded him/ her to continue with monitoring.
  Interventions: Device: Telemonitoring assisted self-care
- Control group (No Intervention): Control group received usual care that includes multidisciplinary care approach in which patients receive guidance and support for self-care. In the care of heart failure (HF) patients, the cardiac team plays a central role in monitoring and interpreting patient symptoms, optimizing medication and providing education. The cardiac team consists of two physicians, one specialized heart failure nurse and a physiotherapist who helps after a hospitalization period. As part of the care process, patients capable of carrying out self-care are identified and they are encouraged to regularly measure their blood pressure, heart rate and weight at home. So far, the information exchange between heart failure patients and care personnel has taken place during patients' visits to the clinic and by telephone. Systematic collection and exploitation of the self-measurement data has been difficult, since it depends on the patient's own activity

INTERVENTIONS:
Device: Telemonitoring assisted self-care — Telemonitoring group was given a home-care package including a weight scale, a blood pressure meter, a mobile phone and self-care instructions. The measurements taken at home to be uploaded were: diastolic and systolic blood pressure, pulse, body weight and an assessment of symptoms. The symptom assessment concerned the patient's feelings of dizziness, dyspnea, palpitation, weakness and, oedema. Patients were also asked to evaluate their overall condition- whether their condition had deteriorated, improved or remained unchanged. The patients were advised to carry out and report the measurements together with the self-assessment once a week. The responsible nurse followed patients' status and the data once a week or more frequently if needed. Based on the reported measurements, the nurse could invite the patient for a control visit. In case a patient did not make self-measurements as planned , the nurse contacted the patient and reminded him/ her to continue with monitoring
  Arms: Telemonitoring assisted self-care

SUMMARY:
In the study benefits of using mobile phone assisted remote patient monitoring including self-measurements of blood pressure, heart rate and weight as well as monitoring of personal health status are investigated in the care of heart failure patients.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of systolic heart failure
* NYHA (New York Heart Association) classification > 1
* left ventricular ejection fraction ≤ 35%
* need for a regular control visit
* time from the last visit no longer than 6 months

Exclusion Criteria:

* Patients who were known to enter a major medical operation
* severe comorbidity,
* participation in other clinical trial during last three months-
* poor compliance in terms of familiarity with mobile phone

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2010-10; Primary Completion 2012-03 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- VTT Technical Research Centre of Finland, Espoo, Finland

REFERENCES:
- [Derived] Vuorinen AL, Leppanen J, Kaijanranta H, Kulju M, Helio T, van Gils M, Lahteenmaki J. Use of home telemonitoring to support multidisciplinary care of heart failure patients in Finland: randomized controlled trial. J Med Internet Res. 2014 Dec 11;16(12):e282. doi: 10.2196/jmir.3651. PMID 25498992

RESULTS

PARTICIPANT FLOW:
Groups:
- Control Group: Control group received multidisciplinary care that was standard.
Period: Overall Study
Arm/Group | Telemonitoring Assisted Self-care | Control Group
Started | 47 | 47
Completed | 46 | 47
Not Completed | 1 | 0
Not completed — Lost to Follow-up | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Telemonitoring-assisted Self-care: Telemonitoring group was given a home-care package including a weight scale, a blood pressure meter, a mobile phone and self-care instructions. The measurements taken at home to be uploaded were: diastolic and systolic blood pressure, pulse, body weight and an assessment of symptoms. The symptom assessment concerned the patient's feelings of dizziness, dyspnea, palpitation, weakness and, oedema. Patients were also asked to evaluate their overall condition- whether their condition had deteriorated, improved or remained unchanged. The patients were advised to carry out and report the measurements together with the self-assessment once a week. The responsible nurse followed patients' status and the data once a week or more frequently if needed. Based on the reported measurements, the nurse could invite the patient for a control visit. In case a patient did not mak
- Control Group: Control group received usual care that includes multidisciplinary care approach in which patients receive guidance and support for self-care. In the care of HF patients, the cardiac team plays a central role in monitoring and interpreting patient symptoms, optimizing medication and providing education. The cardiac team consists of two physicians, one specialized heart failure nurse and a physiotherapist who helps after a hospitalization period. As part of the care process, patients capable of carrying out self-care are identified and they are encouraged to regularly measure their blood pressure, heart rate and weight at home. So far, the information exchange between heart failure patients and care personnel has taken place during patients' visits to the clinic and by telephone. Systematic collection and exploitation of the self-measurement data has been difficult, since it depends on the patient's own activity.
- Total: Total of all reporting groups
Arm/Group | Telemonitoring-assisted Self-care | Control Group | Total
Number analyzed (Participants) | 47 | 47 | 94
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.9 (11.9) | 58.3 (11.6) | 58.0 (11.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 8 | 16
  Male | 39 | 39 | 78
left ventricular ejection fraction [Mean (Standard Deviation); unit: percentage] | 27.3 (4.9) | 28.6 (5.0) | 28.0 (5.0)
NYHA ( Functional Classification of the New York Heart Association) [Number; unit: participants]
  'Slight limitations in physical activity class II' | 19 | 17 | 36
  'Marked limitation in physical activity class III | 27 | 28 | 55
  'Severe limitations in physical activity class IV | 1 | 2 | 3
Body mass index [Mean (Standard Deviation); unit: kg/m2] | 28.4 (6.0) | 27.9 (4.0) | 28.2 (5.4)
Smoking [Number; unit: participants]
  Smoker | 35 | 42 | 77
  Non-smoker | 12 | 5 | 17
Systolic blood pressure [Mean (Standard Deviation); unit: mmHg] | 112 (13) | 116 (16) | 114 (15)
Diastolic blood pressure [Mean (Standard Deviation); unit: mmHg] | 71 (10) | 72 (10) | 72 (10)
NT-proBNP [Median (Inter-Quartile Range); unit: ng/l] — Plasma concentration of brain natriuretic peptide propeptide
  ng/l | 2347 [998 to 3568] | 1338 [474 to 2974] | 1700 [727 to 3433]

OUTCOME MEASURES:

1. Primary Outcome: Number of HF-related Hospital Days
Description: Number of heart failure related hospital days
Time Frame: From baseline until the end of the study at six months
Measure: Mean (Standard Deviation); unit: number of days
Groups:
- Telemonitoring Assisted Self-care: Telemonitoring assisted self-care group was given a home-care package including a weight scale, a blood pressure meter, a mobile phone and self-care instructions. A pre-installed software application in the mobile phone supported uploading of measurements and self-assessment of symptoms. The patients were advised to carry out and report the measurements together with the self-assessment once a week.
  Telemonitoring assisted self-care: The responsible nurse followed patients' status and the data once a week or more frequently if needed. Based on the reported measurements, the nurse could invite the patient for a control visit. In case a patient did not make self-measurements as planned , the nurse contacted the patient and reminded him/ her to continue with monitoring.
- Control Group: Control group received usual care
Arm/Group | Telemonitoring Assisted Self-care | Control Group
Number analyzed (Participants) | 46 | 47
number of days | 0.7 (2.4) | 1.4 (3.5)

2. Secondary Outcome: Death
Description: Death from any cause
Time Frame: From baseline until the end of the study at six months
Measure: Number; unit: participants
Arm/Group | Telemonitoring Assisted Self-care | Control Group
Number analyzed (Participants) | 46 | 47
participants | 0 | 0

3. Secondary Outcome: Heart Transplant
Description: Heart transplant operation or listing for transplant operation
Time Frame: From baseline until the end of the study at six months
Measure: Number; unit: participants
Arm/Group | Telemonitoring Assisted Self-care | Control Group
Number analyzed (Participants) | 46 | 47
participants | 0 | 0

4. Secondary Outcome: P-proBNP
Description: Change in plasma concentration of brain natriuretic peptide propeptide from baseline to the end of the study.
Time Frame: From baseline until the end of the study at six months
Measure: Median (Inter-Quartile Range); unit: ng/l
Arm/Group | Telemonitoring Assisted Self-care | Control Group
Number analyzed (Participants) | 46 | 47
ng/l | -198 [-1921 to 170] | -50 [-831 to 260]

5. Secondary Outcome: EHFSBS (European Heart Failure Self-Care Behaviour Scale ) Scores
Description: Change in self-care behaviour measured by the European Heart Failure Self-Care Behaviour Scale (EHFSBS). EHFSBS is a 12-item self-administered questionnaire specifically designed and tested for heart failure patients including statements on self-care behaviour essential in the care of HF. The statements are scored from one to five. The lower the score, the better the performance in self-care. The summary score is analysed.
Time Frame: From baseline until the end of the study at six months
Measure: Mean (95% Confidence Interval); unit: Scores on a scale
Arm/Group | Telemonitoring Assisted Self-care | Control Group
Number analyzed (Participants) | 46 | 47
Scores on a scale | -5.0 [-7.3 to -3.0] | -3.8 [-5.4 to -2.1]

6. Other Pre Specified Outcome: Plasma Concentrations of Creatinine, Natrium, and Potassium From the Baseline to the End of the Study
Description: Change in plasma concentrations of creatinine, natrium, and potassium
Time Frame: From baseline to the end of the study at six months
Reporting Status: Not Posted

7. Secondary Outcome: Left Ventricular Ejection Fraction
Description: Change in left ventricular ejection fraction from baseline until the end of the study
Time Frame: From baseline until the end of the study at six months
Measure: Mean (95% Confidence Interval); unit: percentage unit
Arm/Group | Telemonitoring Assisted Self-care | Control Group
Number analyzed (Participants) | 46 | 47
percentage unit | 5.0 [1.8 to 8.1] | 4.2 [1.8 to 6.5]

8. Secondary Outcome: Utilization of Health Care Resources
Description: Number of visits to nurse's reception
Time Frame: From baseline until the end of the study at six months
Measure: Mean (Standard Deviation); unit: number of visits
Arm/Group | Telemonitoring Assisted Self-care | Control Group
Number analyzed (Participants) | 46 | 47
number of visits | 4.5 (2.2) | 2.7 (1.0)

ADVERSE EVENTS:
Arm/Group | Telemonitoring Assisted Self-care | Control Group
Serious Adverse Events (participants affected / at risk) | 0/46 | 0/47
Other Adverse Events (participants affected / at risk) | 0/46 | 0/47

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No